CLINICAL TRIAL: NCT07281872
Title: A Single-Center, Randomized, Open-Label, Two-Period, Two-Sequence, Single-Dose, Crossover Bioequivalence Study of Methylconalamin Injection and Methylconalamin for Injection in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of WP205 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: WBD-JGAZSY-I02
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Therapeutic Equivalency, Healthy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Methylconalamin Injection(WP205); Drug: Methylconalamin for Injection
- Group B (Active Comparator)
  Interventions: Drug: Methylconalamin Injection(WP205); Drug: Methylconalamin for Injection

INTERVENTIONS:
Drug: Methylconalamin Injection(WP205) — 25 mg intramuscular injection in the upper-arm deltoid
Drug: Methylconalamin for Injection — 25 mg intramuscular injection in the upper-arm deltoid

SUMMARY:
This study is a single-center, randomized, open-label, two-period, two-sequence, single-dose, crossover bioequivalence trial conducted under fasting conditions in healthy adult volunteers. Participants will be randomized into two sequences (A and B). Each participant will receive a single intramuscular dose of the test or reference formulation according to the assigned sequence, with an adequate washout period between dosing. The primary objective of the study is to evaluate the bioequivalence of the two formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have been fully informed of the study purpose, nature, procedures, and potential adverse reactions, voluntarily agree to participate, and have signed the informed consent form prior to any study-related procedures.
2. Male or female subjects aged 18 years or older, with an appropriate gender distribution.
3. Body weight: females ≥ 45.0 kg, males ≥ 50.0 kg, and body mass index (BMI) between 19.0 and 26.0 kg/m² (inclusive); BMI = weight (kg) / height² (m²).
4. Subjects are able to communicate effectively with the investigators and can understand and comply with all study requirements.

Exclusion Criteria:

1. Known allergy to methylconalamin injection, methylconalamin injection, or any component of the formulations, or history of hypersensitivity (e.g., rash, urticaria).
2. History of clinically significant diseases or any other medical or physiological condition that could interfere with study results, including but not limited to disorders of the hematologic, cardiovascular, digestive, urinary, respiratory, nervous, immune, or endocrine systems, malignancy, psychiatric disorders, or metabolic abnormalities.
3. History of significant bleeding tendency, coagulation disorders, systemic bleeding, neutropenia, or thrombocytopenia.
4. Vaccination with any vaccine or live attenuated vaccine within 1 month prior to dosing, or planned vaccination during the study.
5. Consumption within 48 hours prior to dosing of foods or beverages that may affect metabolism (e.g., grapefruit, pomelo, mango, orange), alcohol, purine-rich or caffeine-containing foods/beverages (e.g., coffee, strong tea, chocolate), or foods rich in vitamin B12 (e.g., animal liver such as pork, beef, chicken, and shellfish such as oysters or clams).
6. Daily excessive consumption of tea, coffee, and/or caffeine-containing beverages (≥8 cups per day, 1 cup = 250 mL) within 3 months prior to screening.
7. Use of any drugs that affect liver enzyme activity within 30 days prior to first dose (e.g., enzyme inducers such as barbiturates, carbamazepine, phenytoin, dexamethasone; inhibitors such as SSRIs, ciprofloxacin, diltiazem, macrolides, metronidazole, ketoconazole, verapamil, fluoroquinolones).
8. Use of any medication (prescription, over-the-counter, herbal, vitamin, or dietary supplement) within 2 weeks prior to screening, except for topical medications or eye drops with local effects.
9. Weekly alcohol consumption exceeding 14 units within 3 months prior to screening (1 unit ≈ 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or positive alcohol breath test, or inability to abstain from alcohol during the study.
10. Smoking ≥5 cigarettes/day within 3 months prior to screening, or inability to stop tobacco use during the study, or positive nicotine test.
11. History of substance abuse within 3 months prior to screening, or positive drug screening.
12. Blood donation or significant blood loss (≥400 mL), transfusion, or use of blood products within 3 months prior to screening, or planned blood donation during the study or within 3 months after study completion.
13. History of surgery within 3 months prior to screening, planned surgery during the study, or history of surgery that may affect drug absorption, distribution, metabolism, or excretion.
14. Use of any investigational drug or participation in any drug/device clinical trial within 1 months prior to screening.
15. Clinically significant abnormalities in vital signs, physical examination, laboratory tests (hematology, urinalysis, blood biochemistry, coagulation), chest X-ray, or 12-lead ECG.
16. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), syphilis antibody (anti-TP), or HIV antibody (anti-HIV).
17. Subjects with special dietary requirements unable to comply with standardized study diet.
18. Subjects unable to tolerate venipuncture or with difficult venous access, or history of orthostatic hypotension, syncope, or needle phobia.
19. Male (or their partner) or female subjects planning pregnancy, egg/sperm donation, unwilling to use effective contraception, positive pregnancy test, or lactating females from signing consent to 1 month after last dose.
20. Subjects deemed unsuitable for participation by their own reason or at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2028-11-25 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0 to 24 hours after each single intramuscular dose
Area under the plasma concentration versus time curve (AUC)0-t | 0 to 24 hours after each single intramuscular dose
Area under the plasma concentration versus time curve (AUC)0-∞ | 0 to 24 hours after each single intramuscular dose

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China